CLINICAL TRIAL: NCT05350657
Title: Ketogenic Dietary Patterns in Young Adults and Kidney Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Sibylle Kranz, PhD, RDN, Associate Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSR210490
Record Dates: First submitted 2021-12-09; First posted 2022-04-28 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Ketogenic Diet; Kidney Injury
Keywords: ketogenic diet; kidney injury
MeSH Terms: interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet (Experimental): Subjects will be provided with foods following a ketogenic diet for 15 consecutive days.
  Interventions: Behavioral: Ketogenic Diet

INTERVENTIONS:
Behavioral: Ketogenic Diet — 2 week isocaloric, high protein and low carbohydrate ketogenic diet

SUMMARY:
This study seeks to assess the kidney health effects of short-term healthful ketogenic diet in young, overweight adults.10 overweight (BMI 25-30 kg/m2) adult participants (ages 20-40 years) without major chronic conditions including diabetes, kidney, cardiac, or liver disease will receive an isocaloric, high protein and low carbohydrate ketogenic diet for 2 weeks.

DETAILED DESCRIPTION:
After baseline measures are taken, 10 overweight (BMI 25-30 kg/m2) young adult participants (ages 20-40 years) without major chronic conditions including diabetes, kidney, cardiac, or liver disease will receive an isocaloric, high protein and low carbohydrate ketogenic diet for 2 weeks. Each participant will consume one meal daily in the Diet and Nutrition (DAN) laboratory metabolic kitchen at the University of Virginia (UVA) and receive the remainder of the daily food allocation packed out to consume at home. Plate-waste method and NDS-R software will be used to measure food consumption (all served and packed-out foods and all uneaten and returned portions will be weighed). Weight, blood pressure and symptom surveys will be monitored at least 3 times a week. Fasting blood and 24 hour urine samples will performed at baseline and the end of each week. Stool for microbiota will be assess at baseline and end of study. Adherence will be confirmed with urinary biomarkers (e.g. urinary nitrogen) and point of care blood testing ketones. Differences in estimated glomerular filtration rate (GFR) determined from serum creatinine and cystatin C will be evaluated for each participant to assess magnitude of increase in GFR on the ketogenic diet. Over the past decade new panels of biomarkers have become available measuring glomerular permeability (urine albumin to creatinine ratio; UACR) and kidney injury and repair (IL-18, kidney injury molecule 1 [KIM-1], neutrophil gelatinase-associated lipocalin [NGAL], liver fatty acid type binding protein [L-FABP], tumor necrosis factor α [TNF-α, TNF receptor 1 and 2], transforming growth factor beta [TGF-β], human cartilage glycoprotein 39 [YKL-40], and monocyte chemoattractant protein 1 [MCP-1]). Change in UACR comparing the end of two weeks to baseline will be the primary outcome. Changes in other kidney injury markers will be assessed as secondary and exploratory outcomes. Additional exploratory outcomes will include urine metabolomics and stool 16S rRNA to characterize the gastrointestinal microbiota. Biosamples will be stored in a repository for future uses.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (BMI 25-30 kg/m2)
* Weight stable for last 4 weeks by self-report
* Residing in the greater Charlottesville/Albemarle area for >6 months out of the last year
* Normal kidney function at baseline, eGFR ≥60 ml/min/1.73m2 and UACR <30 mg/g at screening

Exclusion Criteria:

* History of major medical comorbidities by self-report (history of diabetes; diagnosed kidney disease; diagnosed gastrointestinal disorders including inflammatory bowel disease, gastric bypass, intestinal resection, celiac disease or other malabsorption; esophageal or other disorders limiting ability to swallow food)
* Systolic blood pressure >160 or <100 at screening
* Daily use of diuretics such as hydrochlorothiazide
* Serum potassium <3.5 or >5.1 mEq/L at screening
* Serum magnesium <1.6 mg/dL at screening
* Serum sodium <135 or >149 mEq/L at screening
* HbA1c > 6.5% at screening
* Fasting plasma glucose > 126 mg/dL at screening
* Pregnant or breastfeeding women (confirmed by spot urine at screening)
* Inability to give written informed consent in English
* Inability to walk up to 1 mile at a slow pace between buildings for study visits
* Food allergies
* Eating ketogenic or low carbohydrate diet over last 4 weeks
* Blood ketones positive at screening
* Intolerance or dislike of any study foods limiting adherence
* Inability to attend daily visits
* Vulnerable population such as direct reports or students of the investigators
* Lack of access to refrigeration or equipment to safely reheat meals

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Within-person change in UACR comparing Day 15 to pre-intervention | Day 0 and day 15 of the intervention
  Urine Albumin-Creatinine Ratio comparison tested at alpha 0.05

SECONDARY OUTCOMES:
Within-person change in eGFR-Cr comparing Day 15 to pre-intervention | Day 0 and day 15 of the intervention
  Tested at alpha 0.0125, corrected (Bonferroni correction) for 4 overall outcomes. Due to very high correlation between different eGFR equations these are not corrected as independent tests
Within-person change in eGFR-Cystatin comparing Day 15 to pre-intervention | Day 0 and day 15 of the intervention
  Tested at alpha 0.0125, corrected (Bonferroni correction) for 4 overall outcomes. Due to very high correlation between different eGFR equations these are not corrected as independent tests
Within-person change in eGFR-Cr-and-Cystatin comparing Day 15 to pre-intervention | Day 0 and day 15 of the intervention
  Tested at alpha 0.0125, corrected (Bonferroni correction) for 4 overall outcomes. Due to very high correlation between different eGFR equations these are not corrected as independent tests
Within-person change in urine KIM-1 comparing Day 15 to pre-intervention | Day 0 and day 15 of the intervention
  Tested at alpha 0.0125, corrected (Bonferroni correction) for 4 overall outcomes. Due to very high correlation between different eGFR equations these are not corrected as independent tests
Within-person change in urine NGAL comparing Day 15 to pre-intervention | Day 0 and day 15 of the intervention
  Tested at alpha 0.0125, corrected (Bonferroni correction) for 4 overall outcomes. Due to very high correlation between different eGFR equations these are not corrected as independent tests

OTHER OUTCOMES:
Within-person change in MCP-1 comparing Day 15 to pre-intervention | Day 0 and day 15 of the intervention
  Exploratory and tested at nominal and false discovery rate (FDR)-adjusted p-values
Within person change in urine metabolites comparing Day 15 to pre-intervention | Day 0 and day 15 of the intervention
  Exploratory and tested at nominal and false discovery rate (FDR)-adjusted p-values
Within person change in microbiome composition by 16s rRNA sequencing comparing Day 15 to pre-intervention | Day 0 and day 15 of the intervention
  Exploratory and tested at nominal and false discovery rate (FDR)-adjusted p-values

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Kranz, PhD RDN FTOS, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Buren J, Ericsson M, Damasceno NRT, Sjodin A. A Ketogenic Low-Carbohydrate High-Fat Diet Increases LDL Cholesterol in Healthy, Young, Normal-Weight Women: A Randomized Controlled Feeding Trial. Nutrients. 2021 Mar 2;13(3):814. doi: 10.3390/nu13030814. PMID 33801247
- [Background] Cao J, Lei S, Wang X, Cheng S. The Effect of a Ketogenic Low-Carbohydrate, High-Fat Diet on Aerobic Capacity and Exercise Performance in Endurance Athletes: A Systematic Review and Meta-Analysis. Nutrients. 2021 Aug 23;13(8):2896. doi: 10.3390/nu13082896. PMID 34445057
- [Background] Yancy WS Jr, Westman EC, McDuffie JR, Grambow SC, Jeffreys AS, Bolton J, Chalecki A, Oddone EZ. A randomized trial of a low-carbohydrate diet vs orlistat plus a low-fat diet for weight loss. Arch Intern Med. 2010 Jan 25;170(2):136-45. doi: 10.1001/archinternmed.2009.492. PMID 20101008
- [Background] Hall KD, Guo J, Courville AB, Boring J, Brychta R, Chen KY, Darcey V, Forde CG, Gharib AM, Gallagher I, Howard R, Joseph PV, Milley L, Ouwerkerk R, Raisinger K, Rozga I, Schick A, Stagliano M, Torres S, Walter M, Walter P, Yang S, Chung ST. Effect of a plant-based, low-fat diet versus an animal-based, ketogenic diet on ad libitum energy intake. Nat Med. 2021 Feb;27(2):344-353. doi: 10.1038/s41591-020-01209-1. Epub 2021 Jan 21. PMID 33479499
- [Background] Ludwig DS, Willett WC, Volek JS, Neuhouser ML. Dietary fat: From foe to friend? Science. 2018 Nov 16;362(6416):764-770. doi: 10.1126/science.aau2096. PMID 30442800
- [Background] Mitchell NS, Scialla JJ, Yancy WS Jr. Are low-carbohydrate diets safe in diabetic and nondiabetic chronic kidney disease? Ann N Y Acad Sci. 2020 Feb;1461(1):25-36. doi: 10.1111/nyas.13997. Epub 2019 Jan 15. PMID 30644556
- [Background] Bostock ECS, Kirkby KC, Taylor BV, Hawrelak JA. Consumer Reports of "Keto Flu" Associated With the Ketogenic Diet. Front Nutr. 2020 Mar 13;7:20. doi: 10.3389/fnut.2020.00020. eCollection 2020. PMID 32232045